CLINICAL TRIAL: NCT04367883
Title: Evaluation of Influenza Vaccination and Treatment With ACEI and ARB in the Evolution of SARS-CoV2 Infection
Brief Title: Influenza Vaccination, ACEI and ARB in the Evolution of SARS-CoV2 Infection
Status: Recruiting | Type: Observational
Sponsor: Consorci Sanitari de Terrassa (Other)
Collaborators: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other); Institut Català de la Salut (Other)
Responsible Party: Principal Investigator, Anna Puigdellívol-Sánchez, M.D., Ph.D., Consorci Sanitari de Terrassa
Other Study IDs: 02-20-161-021; 02-22-161-060 (Registry Identifier: Idem + antihistamines, amantadine in the evolution of COVID)
Record Dates: First submitted 2020-04-28; First posted 2020-04-29 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: COVID19; Influenza Vaccination; ACE Inhibitors; ARB; Antihistamine Allergy; Amantadine
MeSH Terms: conditions — COVID-19; Influenza, Human | interventions — Histamine Antagonists; Amantadine; Angiotensin-Converting Enzyme Inhibitors; Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Hospital admissions, postcovid syndrome and thrombosis among COVID cases in CST population: Observation of patient characteristics of hospital incomes in Hospital of Terrassa from March 1, 2020.
  No intervention is performed.
  Interventions: Drug: Antihistamine; Drug: Amantadine; Drug: ACEI; Drug: ARB; Other: Influenza vaccine and COVID
- Evolution of COVID cases in patients receiving antihistamines: COVID cases, hospital admissions, postcovid syndrome, thrombosis and deaths related to COVID from march 1, 2020 in patients of the participating institutions receiving chronic treatment with antihistamines.
  No intervention is performed.
  Interventions: Drug: Antihistamine
- Evolution of COVID cases in patients receiving amantadine.: COVID cases, hospital admissions, postcovid syndrome, thrombosis and deaths related to COVID from march 1, 2020 in patients of the participating institutions receiving chronic treatment with amantadine.
  No intervention is performed.
  Interventions: Drug: Amantadine

INTERVENTIONS:
Drug: Antihistamine — No intervention is performed. We propose an observational study.
  Other Names: Antihistamines for COVID
  Groups: Evolution of COVID cases in patients receiving antihistamines; Hospital admissions, postcovid syndrome and thrombosis among COVID cases in CST population
Drug: Amantadine — No intervention is performed. We propose an observational study
  Other Names: Amantadine for COVID
  Groups: Evolution of COVID cases in patients receiving amantadine.; Hospital admissions, postcovid syndrome and thrombosis among COVID cases in CST population
Drug: ACEI — No intervention is performed. We propose an observational study.
  Other Names: ACEI and COVID
  Groups: Hospital admissions, postcovid syndrome and thrombosis among COVID cases in CST population
Drug: ARB — No intervention is performed. We propose an observational study.
  Other Names: ARB and COVID
  Groups: Hospital admissions, postcovid syndrome and thrombosis among COVID cases in CST population
Other: Influenza vaccine and COVID — No intervention is performed. We propose an observational study.
  Groups: Hospital admissions, postcovid syndrome and thrombosis among COVID cases in CST population

SUMMARY:
Some authors have proposed the use of the flu vaccine to reduce the severity of COVID-19 cases, while some have proposed the use of ACE Inhibitors (ACEI) or Angiotensin Receptor blockers (ARB), since this virus shares hemagglutinin as a transmission mechanism and acts on the ACE2 enzyme during infection.

Other authors described how none of the elderly patients receiving antihistamines and azythromycin in two nursing homes in Toledo -Spain- during the first wave died or needed hospital admission, even considering that 100% of residents had a positive serological test after that wave. Other authors have described a positive evolution in patients receiving amantadine for their Parkinson's disease.

The aim is to evaluate whether the admitted patients who are previously vaccinated or those who were already receiving these treatments showed a better evolution.

DETAILED DESCRIPTION:
The number COVID cases would be related to hospital admissions. Among hospital admissions, the number of previous treatments, the length of admission, the need or not of the Intensive Care Unit (ICU) and their final status (survivors or non survivors) would be studied.

If patients that previously received the influenza vaccine or treated with ACEI, ARB, antihistamines or amantadine showed a better evolution, it would be proposed to extend vaccination and the inclusion of ACE inhibitors, ARB, antihistamines or amantadine in the treatment of infection.

ELIGIBILITY:
Inclusion Criteria:

* Hospital Admissions at the Hospital of Terrassa from March 1, 2020 for any cause.

Exclusion Criteria:

* None.
* For comparison of percentage of Influenza vaccination, ACEI and ARB vs general population, patients from outside the reference area of the Terrassa Health Consortium would be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All hospital admissions in the Hospital of Terrassa from March 1, 2020 were innitially included.
  Population of reference: the population assigned to the Terrassa Health Consortium population.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2025-01-19 (Actual); Study Completion 2028-02-24 (Estimated)

PRIMARY OUTCOMES:
hospital output | from March 1, 2020.
  exitus vs hospital output

SECONDARY OUTCOMES:
hospital stay | From March 1, 2020.
  length of the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Anna Puigdellívol-Sánchez, Ph D, Principal Investigator — Consorci Sanitari de Terrassa
Locations (1):
- Hospital de Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang L, Liu Y. Potential interventions for novel coronavirus in China: A systematic review. J Med Virol. 2020 May;92(5):479-490. doi: 10.1002/jmv.25707. Epub 2020 Mar 3. PMID 32052466
- [Background] Gurwitz D. Angiotensin receptor blockers as tentative SARS-CoV-2 therapeutics. Drug Dev Res. 2020 Aug;81(5):537-540. doi: 10.1002/ddr.21656. Epub 2020 Mar 4. PMID 32129518
- [Background] Moran Blanco JI, Alvarenga Bonilla JA, Homma S, Suzuki K, Fremont-Smith P, Villar Gomez de Las Heras K. Antihistamines and azithromycin as a treatment for COVID-19 on primary health care - A retrospective observational study in elderly patients. Pulm Pharmacol Ther. 2021 Apr;67:101989. doi: 10.1016/j.pupt.2021.101989. Epub 2021 Jan 16. PMID 33465426
- [Background] Cortes-Borra A, Aranda-Abreu GE. Amantadine in the prevention of clinical symptoms caused by SARS-CoV-2. Pharmacol Rep. 2021 Jun;73(3):962-965. doi: 10.1007/s43440-021-00231-5. Epub 2021 Feb 18. PMID 33604795
- [Result] Puigdellivol-Sanchez A, Juanes-Gonzalez M, Calderon-Valdiviezo A, Valls-Foix R, Gonzalez-Salvador M, Lozano-Paz C, Vidal-Alaball J. COVID-19 in Relation to Polypharmacy and Immunization (2020-2024). Viruses. 2024 Sep 27;16(10):1533. doi: 10.3390/v16101533. PMID 39459868
- [Result] Puigdellivol-Sanchez A, Juanes-Gonzalez M, Calderon-Valdiviezo A, Losa-Puig H, Valls-Foix R, Gonzalez-Salvador M, Lozano-Paz C, Vidal-Alaball J. COVID-19 in Relation to Chronic Antihistamine Prescription. Microorganisms. 2024 Dec 13;12(12):2589. doi: 10.3390/microorganisms12122589. PMID 39770791